CLINICAL TRIAL: NCT00231712
Title: Prospective Analysis of the Patterns of Immune Reconstitution Following Conventional or High-Dose Chemotherapy With Autologous/Allogeneic Stem Cell Transplant
Brief Title: Immuno 1: Immune Reconstitution Following Conventional or High-Dose Chemotherapy With Stem Cell Transplant
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Julius-Maximilians University (Other)
Collaborators: University of Wuerzburg (Other)
Other Study IDs: 133/04
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2006-08-23 (Estimated); Status verified 2005-09

CONDITIONS: Leukemia; Medulloblastoma
Keywords: prospective analysis of immune function,; spectratype; immunoscope; TREC analysis; solid tumor
MeSH Terms: conditions — Leukemia; Medulloblastoma

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to conduct an analysis of the influences of

1. conventional chemotherapy
2. high-dose chemotherapy followed by autologous stem cell transplant
3. high-dose chemotherapy followed by allogeneic stem cell transplant on the recovery of the immune system.

Detailed analysis will help to better understand the pathways of recovery of the immune system following chemotherapy as well as the pathways of recovery of the immune system following autologous or allogeneic stem cell transplantation.

DETAILED DESCRIPTION:
Detailed analysis will be performed at preselected time points following therapy by

* standard flow cytometry in combination with intracellular cytokine/antigen staining
* spectratype analysis
* TREC assays

ELIGIBILITY:
Inclusion Criteria:

* Acute leukemia treated according to current ALL-BFM 2002 protocol
* Solid tumor treated according to current GPOH-protocol
* Medulloblastoma treated according to HIT-2000 protocol
* High-dose chemotherapy followed by autologous stem cell transplantation
* High-dose chemotherapy followed by allogeneic stem cell transplantation
* Written consent according to our institutional guidelines

Exclusion Criteria:

* No written consent

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2005-03; Study Completion 2009-02

CONTACTS AND LOCATIONS:
Overall Officials: Paul G Schlegel, MD, Principal Investigator — University Children's Hospital Pediatric Oncology Wuerzburg / Germany; Matthias Eyrich, MD, Study Director — Pediatric Stem Cell Transplant Program
Locations (1):
- University Children's Hospital Pedaitric Oncology, Würzburg, Germany

REFERENCES:
- [Background] Eyrich M, Wollny G, Tzaribaschev N, Dietz K, Brugger D, Bader P, Lang P, Schilbach K, Winkler B, Niethammer D, Schlegel PG. Onset of thymic recovery and plateau of thymic output are differentially regulated after stem cell transplantation in children. Biol Blood Marrow Transplant. 2005 Mar;11(3):194-205. doi: 10.1016/j.bbmt.2004.12.001. PMID 15744238
- [Background] Eyrich M, Leiler C, Lang P, Schilbach K, Schumm M, Bader P, Greil J, Klingebiel T, Handgretinger R, Niethammer D, Schlegel PG. A prospective comparison of immune reconstitution in pediatric recipients of positively selected CD34+ peripheral blood stem cells from unrelated donors vs recipients of unmanipulated bone marrow from related donors. Bone Marrow Transplant. 2003 Aug;32(4):379-90. doi: 10.1038/sj.bmt.1704158. PMID 12900774
- [Background] Eyrich M, Croner T, Leiler C, Lang P, Bader P, Klingebiel T, Niethammer D, Schlegel PG. Distinct contributions of CD4(+) and CD8(+) naive and memory T-cell subsets to overall T-cell-receptor repertoire complexity following transplantation of T-cell-depleted CD34-selected hematopoietic progenitor cells from unrelated donors. Blood. 2002 Sep 1;100(5):1915-8. doi: 10.1182/blood-2001-11-0005. PMID 12176918